CLINICAL TRIAL: NCT05239858
Title: International Wilson's Disease Patient Registry (iWilson Registry)
Status: Recruiting | Type: Observational
Sponsor: Orphalan (Industry)
Collaborators: Ergomed (Industry)
Responsible Party: Sponsor
Other Study IDs: ORPH-131-005
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Wilson's Disease
Keywords: trientine; d-Penicillamine; ATP7B; hepatolenticular degeneration; copper metabolism; zinc
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Longitudinal, observational, non-interventional, standard of care Registry. Data will be collected from the routinely scheduled WD clinic visits at approximately 6-12 month intervals. At enrolment, in addition to data from the clinic visit, retrospective data will be collected from the diagnostic evaluation and any relevant past medical history and a summary of WD medication history.

DETAILED DESCRIPTION:
This is a retrospective/prospective observational registry without a control group. A standardised collection tool will be utilised to capture and compare data. The registry will use common data elements, guided by a literature review, and expert input from the multidisciplinary advisory board. The SF-12 Health Survey will be requested from patients aged 18 and over at entry to the Registry to provide a snapshot of baseline quality of life assessment in patients with WD. This will enhance generalisability (external validity) and comparability with clinical trial data.

The objectives of the registry are:

1. Natural history of diagnosis and treated WD patients by documentation of observed clinical practice and patient experience
2. Measure, and compare epidemiological and clinical aspects of Wilson Disease (WD) in the participating countries, thereby encouraging the identification of new standards for the management of WD
3. To provide data for epidemiological research and identify groups of patients potentially eligible for multi-centre trials
4. Describe clinical pathways, by documenting standardised examinations and tests used to monitor WD patients including tools to evaluate adherence and compliance to therapies using real-world outcomes.
5. To be more inclusive (heterogeneous patient population; paediatric, adults, elderly) using much broader inclusion criteria and fewer exclusion criteria than commonly used in randomised trials.
6. Longer follow-up compared to RCTs beneficial detecting delayed or long-term benefits or harm and surveillance for rare events of the disease itself or therapies

Patients will be seen as per their usual standard of care visits. Data points of interest for the Registry will be collected. These may include but not limited to: Medical history, Wilson's Disease Diagnosis and Medical History, Genetics, Liver Assessments, Fibrosis Stage, Liver Transplant, Neurological Assessments, Psychological Assessments, Clinical Global Impression of Change Scale (CGIC), Laboratory measurements incl. Urinary Copper Excretion and Free Copper (NCC), Physical Examination, Adverse Reactions and Serious Adverse Reactions documented by physicians

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide, and has provided, written informed consent/assent
2. Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable, including:

   1. For US sites: Authorization for Use and Release of Health Research Study Information
   2. For EU sites: Data Protection Consent
3. All patients diagnosed with WD including pre-symptomatic individuals and individuals with co-morbidities/diagnoses
4. Any treatments including prescribed and homeopathic/traditional therapies or naive patients on no therapy

Exclusion Criteria:

1. Refusal of informed consent by either patient or their legally acceptable guardian

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Registry aims to be as inclusive as possible. All patients with WD (adult and paediatric ≥12) who provide informed consent/assent can be included. They will be approached during regular follow up visits for ongoing care of their Wilson's Disease by their primary physician.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Describe the natural history of treated WD | 5 years
  Describe the natural history of treated WD and to explore the clinical phenotype, geographic, ethnic and gender influences on the course of the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Mistry, PhD, Study Chair — Yale University Hospital, Conneticut
Locations (16):
- University Hospital Leuven, Leuven, Belgium
- France (2):
  - Hospices Civils de Lyon, Bron, Auvergne-Rhône-Alpes
  - HF Adolphe de Rothschild, Paris, Île-de-France Region
- Germany (4):
  - Charite-Univeritatsmedizin Berlin Hospital, Berlin
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Hannover Medical School (MHH), Hanover
  - Universitätsklinikum Leipzig, Leipzig
- Poland (2):
  - Institute of Psychiatry and Neurology, Warsaw
  - The Children's Memorial Health Institute, Warsaw
- King Faisal Specialist Hospital in Riyadh, Riyāḑ, Riyadh Region, Saudi Arabia
- Spain (4):
  - Hospital Universitario GC Dr Negrín, Las Palmas de Gran Canaria, Canary Islands
  - University Hospital Clínic de Barcelona, C. de Villarroel, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Y Politécnico La Fe, Valencia
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Free Hospital, London